CLINICAL TRIAL: NCT05445323
Title: A Phase 1/2 Study of the Safety and Efficacy of LX2006 Gene Therapy in Participants With Cardiomyopathy Associated With Friedreich's Ataxia
Brief Title: Gene Therapy for Cardiomyopathy Associated With Friedreich's Ataxia
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Lexeo Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LX2006-01
Record Dates: First submitted 2022-06-23; First posted 2022-07-06 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Friedreich Ataxia; Cardiomyopathy, Secondary
Keywords: Friedreich's Ataxia; Cardiomyopathy; FA; Gene therapy; FXN Gene; Frataxin Gene; LX2006
MeSH Terms: conditions — Friedreich Ataxia; Cardiomyopathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cohort 1/ Cohort 2/ Cohort 3 (Experimental)
  Interventions: Genetic: Low dose LX2006; Genetic: Mid Dose LX2006; Genetic: High Dose LX2006

INTERVENTIONS:
Genetic: Low dose LX2006 — Adeno-associated viral vector encoding the FXN gene (AAVrh.10hFXN)
Genetic: Mid Dose LX2006 — Adeno-associated viral vector encoding the FXN gene (AAVrh.10hFXN)
Genetic: High Dose LX2006 — Adeno-associated viral vector encoding the FXN gene (AAVrh.10hFXN)

SUMMARY:
This is a Phase 1/2, open-label, dose-ascending, multicenter study of the safety and efficacy of LX2006 for participants who have Friedreich's Ataxia with evidence of cardiomyopathy. The study will evaluate up to three doses of single administration of LX2006 (AAVrh.10hFXN), an adeno-associated virus (AAV) gene therapy designed to intravenously deliver the human frataxin (hFXN) gene to cardiac cells over a 52-week period. Long-term safety and efficacy will be evaluated for an additional 4-years for a total of 5-years post LX2006 treatment.

DETAILED DESCRIPTION:
Friedreich's ataxia (FA) is a rare, autosomal recessive disease caused by a mutation in the autosomal frataxin (FXN) gene. Progressive cardiomyopathy with cardiac hypertrophy and fibrosis is observed in most individuals with FA. The disease is more severe in those with earlier onset. Presently, there is no therapy that alters the progression of cardiomyopathy in FA, which is responsible for 59% of FA-related deaths.

The primary objective of this dose escalation study is to assess the safety and tolerability of three ascending doses of LX2006 in patients with FA-associated cardiomyopathy. LX2006 is designed to restore hFXN levels in order to improve mitochondrial function. Assessments of cardiac function, biomarkers and other preliminary efficacy endpoints are also included in this study.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed genetic diagnosis of FA, with onset being before 25 years of age
* Protocol specified ranges for antibodies
* Protocol specified measures of FA cardiomyopathy

Exclusion Criteria:

* Protocol specified ranges for left ventricular ejection fraction (LVEF) as measured by cardiac ECHO
* Uncontrolled diabetes
* Abnormal liver function
* Active infection of any type, including hepatitis virus (A, B or C) or human immunodeficiency virus (HIV-1 and HIV-2)
* Contraindication to cardiac MRI
* Contraindications to cardiac biopsies
* Participants who are receiving systemic corticosteroids or other immunosuppressive medications
* History of significant coronary artery disease or any structural heart or vascular disease other than FA cardiomyopathy
* Presence of clinically significant, hemodynamically unstable arrhythmias, requiring physician intervention
* Presence of clinically significant abnormalities as determined by the investigator, other than ECG abnormalities related to FA
* Uncontrolled psychiatric disease

Other Inclusion/Exclusion criteria to be applied as per protocol.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2022-08-24 (Actual); Primary Completion 2029-09 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Treatment-emergent adverse events (TEAEs) and Treatment-emergent serious events (TESAEs) | Change from baseline to end of year 5 post dose

SECONDARY OUTCOMES:
Change from baseline in LVMi | Change from baseline to end of year 5 post dose
Change from baseline in LVEF | Change from baseline to end of year 5 post dose
Change from baseline in cardiac fibrosis as measured by cardiac MRI | Change from baseline to end of year 5 post dose
Change from baseline in measures of cardiopulmonary exercise tolerance | Change from baseline to end of year 5 post dose
Presence and severity of cardiac arrythmias | Change from baseline to end of year 5 post dose

CONTACTS AND LOCATIONS:
Overall Officials: LEXEO Clinical Trials, Study Director — Lexeo Therapeutics
Locations (3):
- United States (3):
  - Ataxia Center and HD Center of Excellence, University of California, Los Angeles, California
  - University of South Florida, Tampa, Florida
  - Mayo Clinic, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No